CLINICAL TRIAL: NCT00318396
Title: Compaction Femur Total Hip Arthroplasty (THA) Uni-lateral
Brief Title: Compaction Femur Preparation for Cementless Total Hip Arthroplasty (THA) Unilateral
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ON-04-002a-SKO
Record Dates: First submitted 2006-04-23; First posted 2006-04-26 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Coxarthrosis
Keywords: THA
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Compaction (Experimental): The bone is pressed very hard together before implantation of femoral component.
  Interventions: Procedure: Bone preparation technique: compaction
- Conventional technique (Active Comparator): The bone is broached before implantation of femoral component.
  Interventions: Procedure: Bone preparation technique: conventional technique

INTERVENTIONS:
Procedure: Bone preparation technique: compaction — The bone is pressed very hard together before implantation of femoral component.
  Other Names: No other names.
  Arms: Compaction
Procedure: Bone preparation technique: conventional technique — Bone is broached before implantation of femoral component.
  Other Names: No other names.
  Arms: Conventional technique

SUMMARY:
This is a prospective, randomized study comparing two different bone preparation techniques for insertion of a hydroxylapatite (HA) coated titanium cementless femoral stem. Patients who receive a unilateral total hip replacement are randomized to either conventional broaching or compaction.

Hypothesis: Compaction results in significantly less stem migration [evaluated by radiostereometric analysis (RSA)], less peri-prosthetic bone mineral density (BMD) loss [evaluated by dual energy x-ray absorptiometry (DEXA)], and a higher Harris hip score after two years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary arthritis in the hip
* Patients with sufficient bone density to allow uncemented implantation of a femoral component
* Informed patient consent in writing

Exclusion Criteria:

* Patients with neuromuscular or vascular disease in the affected leg
* Patients found upon operation to be unsuited for uncemented acetabulum component
* Patients who regularly take non-steroidal anti-inflammatory drugs (NSAIDs) and cannot interrupt intake for the postoperative phase of the study
* Patients with fracture sequelae
* Female patients of childbearing capacity
* Hip joint dysplasia
* Sequelae to previous hip joint disorder in childhood

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2004-06; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
To examine a possible difference in density of bones around implantation of femoral component. | 5 years
  A check-up by means of DEXA scanning after 1 week, 1 year, 2 years and 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Soeren Kold, MD, Principal Investigator — Northern Orthopaedic Division; Kjeld Soeballe, MD, Prof., Study Director — Aarhus University Hospital
Locations (1):
- Northern Orthopaedic Division, Clinic Farsoe, Aalborg University Hospital, Farsø, Northern Jutland, Denmark